CLINICAL TRIAL: NCT06750224
Title: Comparative Effects of Alexander Techniques and Feldenkrais Method on Balance, Fear of Fall and Quality of Life in Patients With Parkinson's Disease.
Brief Title: Comparative Effects of Alexander Techniques and Feldenkrais Method in Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0248
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Alexander techniques; balance; Feldenkrais method; fear of fall; quality of life; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alexander (Experimental): Group A will receive therapy according to Alexander techniques for every alternate day (3 days per week) for 8 weeks. Total 40 minutes of session.
  Interventions: Other: Alexander technique
- feldenkrais (Experimental): Group B will receive therapy according to Feldenkrais method for every alternate day (3 days per week) for 8 weeks. Total 40 minutes of session
  Interventions: Other: Feldenkrais method

INTERVENTIONS:
Other: Alexander technique — 24 sessions for 8 weeks, per week 3 sessions will be given
  Arms: alexander
Other: Feldenkrais method — The method is divided into eight lessons according to 'Awareness Through Movement'. Each lesson will be given three times for one week.
  Arms: feldenkrais

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by tremors, rigidity, and postural instability. These symptoms significantly impact balance and increase the risk of falls, which subsequently lead to a heightened fear of falling and a diminished quality of life. Alexander Technique and the Feldenkrais Method have shown effects in improving overall well-being.

The study is randomized clinical trial will be carried at General hospital. 46 participants meeting the inclusion criteria will be included in this study. Participants will be randomly assigned into 2 groups, Group A and Group B participants will receive Alexander techniques and Feldenkrais method, respectively. All the groups will receive interventions for three days a week for 8 weeks.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by motor symptoms such as tremors, rigidity, bradykinesia, and postural instability. These symptoms significantly impact balance and increase the risk of falls, which subsequently lead to a heightened fear of falling and a diminished quality of life. Alexander Technique and the Feldenkrais Method have shown promise in improving motor function and overall well-being. The primary objective of this study is to compare the effects of the Alexander Technique and the Feldenkrais Method on balance, fear of falling, and quality of life in patients with Parkinson's disease.

This randomized clinical trial will be carried at General hospital after the approval of permission letter. Total number of 46 participants meeting the inclusion criteria will be included in this study through a non-probability convenient sampling technique. Participants will be randomly assigned into 2 groups using computer generated randomization method. Group A and Group B participants will receive Alexander techniques and Feldenkrais method, respectively. All the groups will receive interventions for three days a week for 8 weeks. Total treatment time will be 40 minutes. The outcome measuring scales used will be Berg balance scale and time-up and go to measure balance, fall efficacy scale-international to measure fear of fall, and the Parkinson's disease questionnaire (PDQ-39) to measure quality of life. The data will be collected at baseline and after 8 weeks of therapy, to measure the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* The age group of 50 to 70 years will be included.
* Both genders (male and female)
* Patients diagnosed with Parkinson's disease of Hoehn and Yahr stage (1-3).
* Patient should be able to stand 10 minutes at least without assistance.
* Patients should be able to walk with or without assistance.
* MMSE (score higher than 24).

Exclusion Criteria:

* Recent surgery or any fracture
* Visual and hearing impairments.
* CVS impairments that interfered with therapy
* Joint pain or musculoskeletal problem that interfered with therapy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Berg balance scale | 8 weeks
  It is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait. A score of 56 indicates functional balance. A score of <45 indicates individuals may be at greater risk of falling. A score of ≤49 indicates a risk of falls in individuals with stroke.
Time up and go (TUG) | 8 weeks
  The patient starts in a seated position. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling. In Parkinson's, the patient is at high risk of fall if he takes more than 11.5 seconds.
Fall efficacy scale-international (FES-I) | 8 weeks
  It is a 16-item questionnaire, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Quality of life questionnaire for Parkinson's PDQ-39 | 8 weeks
  PDQ-39 comprises 39 questions from 8 dimensions which include mobility, activities of daily of living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phill, Principal Investigator — Riphah International University
Locations (1):
- General hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teixeira-Machado L, de Araújo FM, Menezes MA, Cunha FA, Menezes T, Ferreira CdS, et al. Feldenkrais method and functionality in Parkinson's disease: a randomized controlled clinical trial. International Journal on Disability and Human Development. 2017;16(1):59-66.
- [Background] Sedaghati P, Goudarzian M, Daneshmandi H, Ardjmand A. Effects of Alexander-based corrective techniques on forward flexed posture, risk of fall, and fear of falling in idiopathic Parkinson's disease. Archives of Neuroscience. 2018;5(2).
- [Background] Hafezi M, Rahemi Z, Ajorpaz NM, Izadi FS. The effect of the Alexander Technique on pain intensity in patients with chronic low back pain: A randomized controlled trial. J Bodyw Mov Ther. 2022 Jan;29:54-59. doi: 10.1016/j.jbmt.2021.09.025. Epub 2021 Oct 9. PMID 35248289
- [Background] Kang SH, Kim J, Kim I, Moon YA, Park S, Koh SB. Dance Intervention Using the Feldenkrais Method Improves Motor, and Non-Motor Symptoms and Gait in Parkinson's Disease: A 12-Month Study. J Mov Disord. 2022 Jan;15(1):53-57. doi: 10.14802/jmd.21086. Epub 2021 Nov 3. PMID 34724780
- [Background] Gross M, Condie C, Grieb J, Cohen R. Poised for Parkinson's: Retention of benefits 6-7 months after Alexander technique synchronous online group course. Archives of Physical Medicine and Rehabilitation. 2022;103(12):e150.
- [Background] Babaei H, Alizadeh MH, Minoonezhad H, Movahed A, Maher R. Effectiveness of the Alexander Technique on quality of life in young men with upper crossed syndrome. Physical Treatments-Specific Physical Therapy Journal. 2024;14(2):125-36.
- [Background] Berland R, Marques-Sule E, Marin-Mateo JL, Moreno-Segura N, Lopez-Ridaura A, Sentandreu-Mano T. Effects of the Feldenkrais Method as a Physiotherapy Tool: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2022 Oct 22;19(21):13734. doi: 10.3390/ijerph192113734. PMID 36360614
- [Background] Pour Kamali T, Yazdkhasti F, Oreyzi HR, Chitsaz A. A Comparison of Effectiveness of Dohsa-hou and the Alexander Technique on Happiness, Social Adjustment, Hope, Mental Health, and Quality of Life in Patients with Parkinson's Disease. Japanese Psychological Research. 2018;60(2):87-98.
- [Background] Cohen RG, Baer JL, Ravichandra R, Kral D, McGowan C, Cacciatore TW. Lighten Up! Postural Instructions Affect Static and Dynamic Balance in Healthy Older Adults. Innov Aging. 2020 Mar 24;4(2):igz056. doi: 10.1093/geroni/igz056. eCollection 2020. PMID 32226825